CLINICAL TRIAL: NCT05943808
Title: Teaching Acupuncture Points With Recorded VR Courses Versus Traditional Text
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH111-REC3-186
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Acupuncture Learning

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Book reading: Test subjects in this group are given a page range within a traditional acupuncture text book to study for 30 minutes.
  Interventions: Other: Book reading
- VR pre-recorded video watching: Test subjects in this group are given a video which was pre-recorded with our Virtual reality system to study for 30 minutes.
  Interventions: Other: VR pre-recorded video watching

INTERVENTIONS:
Other: Book reading — subjects are given an acupuncture textbook to read for 30 minutes
  Groups: Book reading
Other: VR pre-recorded video watching — subjects are given an pre-recorded VR video to watch for 30 minutes
  Groups: VR pre-recorded video watching

SUMMARY:
Compare the learning effectiveness of traditional book learning and VR pre-recorded courses as a reference for future development of VR teaching systems

DETAILED DESCRIPTION:
Traditional Chinese medicine acupuncture education primarily relies on two-dimensional textbooks as the main learning method. Although supplementary materials such as anatomy courses and acupoint anatomy books can partially compensate for the shortcomings of traditional textbooks in anatomical integration, these materials only provide predetermined anatomical views. They make it difficult for students to learn from arbitrary angles and anatomical levels. Therefore, the investigators are developing a Virtual Reality (VR) acupuncture bronze figure model and learning system in an attempt to enhance the depth of acupuncture point learning beyond traditional methods. In this research, the investigators will compare the learning outcomes of traditional book learning and VR pre-recorded courses.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have not previously been exposed to any courses related to Traditional Chinese Medicine acupuncture.
2. Participants who have received an explanation of the research purpose and the entire experimental process, have consented to participate in the study, and have signed an informed consent form.

Exclusion Criteria:

1. Individuals who refuse to sign the informed consent form.
2. The project leader and research advisors.
3. Students who have a direct teaching relationship with the researchers.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mainly bachelor degree students
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Test score change | within singe 1 hour session
  Test subjects are first given a paper exam comprising of 40 questions. Exam time of 15 minutes. Subjects then study based on the assigned group. After 30 minutes of study. Subjects then take another paper exam (15 minutes).

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, North District, Taiwan

IPD SHARING:
Plan to Share IPD: No
There are currently no plans to share data.